CLINICAL TRIAL: NCT01122017
Title: A Modified (Retro-Tubercle) Opening Wedge High Tibial Osteotomy Versus the Conventional Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Dr. Mohammad Reza Abbasian, Department of Orthopedic Surgery, Akhtar Hospital, Shaheed Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBMU-400/435
Record Dates: First submitted 2009-12-01; First posted 2010-05-12 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-04

CONDITIONS: Genu Varum
MeSH Terms: conditions — Genu Varum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medial Opening-Wedge Osteotomy (Experimental): Medial Opening-Wedge Osteotomy (MOWO) is an approach for the correction of malalignment of the knee
  Interventions: Procedure: Retro-Tubercle Opening-Wedge High Tibial Osteotomy

INTERVENTIONS:
Procedure: Retro-Tubercle Opening-Wedge High Tibial Osteotomy — Retro-Tubercle Opening-Wedge High Tibial Osteotomy (ROWHTO) is among the latest approaches for the treatment of varus deformity of knee.

SUMMARY:
The present study was conducted among a group of Iranian patients suffering from varus knee in order to compare advantages and disadvantages of ROWHTO (Retro-Tubercle Opening Wedge High Tibial Osteotomy) technique when compared with previously described approaches of opening-wedge osteotomy.

DETAILED DESCRIPTION:
There are various methods for correcting varus deformity; therefore the best surgical method must be individualized. We concluded that in a varus knee where only correction in the coronal plane without patella infra, changes in Q- angle, tibial plateau inclination is all that is needed, a retro- tubercle medial opening- wedge osteotomy is the preferred approach.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic varus deformity of the knee with 2 or more degrees of anatomical axis varus without ligament injury

Exclusion Criteria:

* fractures through compartments of the knee or the patella
* osteoarthritis other than in the medial compartment
* 10 degrees or more extension lag
* tibial malrotation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-01; Primary Completion 2008-02 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The proportion of patellar length (in mm)to the patellar tendon length (in mm) | up to 13 months
  The length of the patella (in its longest diameter on a lateral x-ray) to the length of the patellar tendon is referred as Insall-Salvati index
The proportion of patellar articular surface length (in mm)to the patella-tibial plateau distance (in mm) | up to 13 months
  The length of the articular surface of the patella to the distance from the patella to the tibial plateau is referred as Blackburne-Peel index.

SECONDARY OUTCOMES:
Quadriceps angle in degree | up to 13 months
  The angle between the quadriceps vector and the line of pull of the patellar tendon from the centre of the patella to the tibial tubercle.
Inclination of proximal tibial plateau in degree | up to 13 months
  The angle between articular surface and lateral longitudinal axis of tibia.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Reza Abbasian, Dr., Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shahid Beheshti University of Medical Sciences, Tehran, Tehran Province, Iran